CLINICAL TRIAL: NCT05165797
Title: Platelet Activation Affecting the Rate of Vascular Access Patency; Single Center, Prospective Observational Study
Brief Title: Platelet Activation Affecting the Rate of Vascular Access Patency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Gwon, Jun Gyo, Associate professor, Korea University Anam Hospital
Other Study IDs: KoreaUAnamH
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Platelet Activation; Hemodialysis Fistula Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: platelet activation factors — platelet activation factors of subject blood

SUMMARY:
In the case of cardiovascular diseases such as coronary artery disease, cerebrovascular disease, and peripheral arterial disease, there are many studies that the use of antiplatelet agents is very helpful in improving the vascular patency rate, but there are not many studies on the use of antiplatelet agents in the dialysis approach. The basis for use is insufficient. There is a lack of research on whether maintaining a state in which platelet activation is suppressed is helpful in improving dialysis access patency. Therefore, we conducted this study to determine whether the degree of platelet activation affects the patency of vascular access.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 years of age or older who are undergoing hemodialysis during renal replacement therapy
* Patients undergoing arteriovenous fistula formation and hemodialysis to the affected area
* Patients who have the ability and willingness to consent to participate in the clinical study, have signed the consent form in accordance with the appropriate procedures, and can visit and participate in the clinical study as planned

Exclusion Criteria:

* Patients who failed to start hemodialysis with an arteriovenous fistula within 3 months
* Patients who have had stent implantation or surgery during the study period due to cardiovascular disease
* Patients with severe hepatic impairment
* Patients with coagulopathy and liver disease associated with clinically significant bleeding risk
* Patients with clinically significant bleeding or bleeding risk
* Patients who underwent artificial heart valve replacement requiring anticoagulant administration
* Patients with pulmonary embolism who are hemodynamically unstable or require thrombolysis or pulmonary embolization.
* Pregnant and lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing dialysis access route formation for the purpose of hemodialysis at this institution
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Vascular access primary patency | 1 month
  Time from vascular access creation until hemodialysis related procedure

SECONDARY OUTCOMES:
Vascular access secondary patency | 1 month
  Time from vascular access creation until hemodialysis failure

CONTACTS AND LOCATIONS:
Locations (1):
- Korea university anam hospital, Seoul, Non US/Canada, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) cannot be shared with other researchers as it is the patient's medical information.